CLINICAL TRIAL: NCT03359291
Title: A Single-center, Open-label, One-sequence, Two-treatment Study to Investigate the Effect of Macitentan at Steady State on the Pharmacokinetics of Rosuvastatin in Healthy Male Subjects.
Brief Title: Clinical Study to Investigate the Effect of Macitentan on the Concentrations of Rosuvastatin in the Blood of Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-055-122
Record Dates: First submitted 2017-11-13; First posted 2017-12-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects
Keywords: macitentan; rosuvastatin; pharmacokinetics
MeSH Terms: interventions — Rosuvastatin Calcium; macitentan

STUDY DESIGN:
Intervention Model Description: All subjects will receive rosuvastatin alone (treatment A) or with macitentan at steady state (treatment B). A fixed sequence design was selected to avoid a lengthy washout period and unnecessary prolongation of subjects' participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence AB (Experimental): Subjects participate in two study periods: During the first period (treatment A), they receive a single oral dose of rosuvastatin on Day 1. During the second period (treatment B), they receive a single oral loading dose of macitentan on Day 5 and oral doses of macitentan from Day 6 to Day 16 (i.e., 11 doses). Subjects receive a single oral dose of 10 mg rosuvastatin concomitantly with macitentan in the morning of Day 10.
  Interventions: Drug: Rosuvastatin; Drug: Macitentan

INTERVENTIONS:
Drug: Rosuvastatin — Single oral dose of 10 mg rosuvastatin (film-coated tablet) on Day 1 and Day 10
Drug: Macitentan — Single oral dose of 30 mg macitentan (film-coated tablet) on Day 5 and 10 mg macitentan administered orally from Day 6 to Day 16
  Other Names: ACT-064992

SUMMARY:
The aim of this Phase 1 trial is to study a potential drug-drug interaction between macitentan and rosuvastatin, a model substrate of various transporter proteins (e.g. in the gut).

DETAILED DESCRIPTION:
Rosuvastatin is a substrate of various transporter proteins including breast cancer resistance protein (BCRP) and organic anion-transporting polypeptides (OATP). It is unknown to which extent macitentan has an effect, if any, on BCRP transporters, especially intestinal BCRP. The primary purpose of this Phase 1 study is to investigate the effect of macitentan on the pharmacokinetics of rosuvastatin, a model BCRP substrate.

ELIGIBILITY:
Principal Inclusion Criteria:

* Signed informed consent in the local language prior to any study-mandated procedure.
* Healthy male subjects aged between 18 and 55 years (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Body mass index of 18.0 to 30.0 kg/m2 (inclusive) at screening.
* Systolic blood pressure 100-140 mmHg, diastolic blood pressure 60-90 mmHg, and pulse rate 50-90 beats per minute (inclusive), measured on the dominant arm, after 5 min in the supine position at screening.
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, measured after 5 min in the supine position at screening.
* Hematology and clinical chemistry test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen and alcohol breath test at screening and Day -1.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Principal Exclusion Criteria:

* Known allergic reactions or hypersensitivity to macitentan, rosuvastatin, any drug of the same classes, or any of their excipients.
* Any contraindication for rosuvastatin treatment.
* History or clinical evidence of myopathy.
* Subjects of Asian race.
* Known hypersensitivity or allergy to natural rubber latex.
* Values of hepatic aminotransferase (alanine aminotransferase and aspartate aminotransferase) outside of the normal range at screening.
* Hemoglobin or hematocrit outside of the normal range at screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study treatment(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Veins unsuitable for intravenous puncture on either arm (e.g., veins that are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture).
* Previous exposure to macitentan.
* Previous exposure to rosuvastatin.
* Treatment with another investigational drug within 3 months prior to screening or participation in more than 3 investigational drug studies within 1 year prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening.
* Nicotine intake (e.g., smoking, nicotine patch, nicotine chewing gum or electronic cigarettes) within 3 months prior to screening and inability to refrain from nicotine intake from screening until End-Of-Study (EOS).
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 3 weeks prior to first study treatment administration.
* Loss of 250 mL or more of blood within 3 months prior to screening.
* Positive results from the hepatitis serology, except for vaccinated subjects or subjects with past but resolved hepatitis, at screening.
* Positive results from the HIV serology at screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) of rosuvastatin following administration of rosuvastatin alone (treatment A) and in combination with macitentan (treatment B) | From Day1 to Day17 (treatment A: from Day1-Day5 and treatment B: from Day10-Day17)
  AUC(0-inf) is the area under the plasma concentration-time curves of rosuvastatin, calculated from time zero to the extrapolated infinite time
Cmax of rosuvastatin following administration of rosuvastatin alone (treatment A) and in combination with macitentan (treatment B) | From Day1 to Day17 (treatment A: from Day1-Day5 and treatment B: from Day10-Day17)
  Cmax is the maximum observed plasma concentration and is directly derived from the individual plasma concentration time curves of rosuvastatin

SECONDARY OUTCOMES:
tmax of rosuvastatin following administration of rosuvastatin alone (treatment A) and in combination with macitentan (treatment B) | From Day1 to Day17 (treatment A: from Day1-Day5 and treatment B: from Day10-Day17)
  The time to reach maximum plasma concentration (tmax) of rosuvastatin
t½ of rosuvastatin following administration of rosuvastatin alone (treatment A) and in combination with macitentan (treatment B) | From Day1 to Day17 (treatment A: from Day1-Day5 and treatment B: from Day10-Day17)
  t½ is the terminal half-life of rosuvastatin and corresponds to the period of time required for the concentration levels of rosuvastatin to be reduced by one-half
AUC(0-t) of rosuvastatin following administration of rosuvastatin alone (treatment A) and in combination with macitentan (treatment B) | From Day1 to Day17 (treatment A: from Day1-Day5 and treatment B: from Day10-Day17)
  AUC(0-t) is the area under the plasma concentration-time curve from time zero to time t of the last measured concentration above the limit of quantification of rosuvastatin
Trough plasma concentrations of macitentan and its metabolite ACT-132577 | From Day5 to Day17
  Trough concentrations of macitentan and ACT-132577 are measured before oral administration of macitentan
Change from baseline in supine blood pressure | From Day1 to end-of-study visit (Day 26-28)
  Change from baseline to each time point of measurement during study period
Change from baseline in pulse rate | From Day1 to end-of-study visit (Day 26-28)
  Change from baseline to each time point of measurement during study period
Change from baseline in heart rate (HR) | From Day1 to end-of-study visit (Day 26-28)
  Change from baseline to each time point of measurement during study period
Change from baseline in ECG variables | From Day1 to end-of-study visit (Day 26-28)
  Change from baseline to each time point of measurement during study period in ECG variables: PR, QRS, QT, RR, and QT corrected for Bazett's and Fridericia's formulae (QTcB and QTcF, respectively)
Change from baseline to end-of-study (EOS) in body weight | From Day1 to end-of-study visit (Day 26-28)
  Change in body weight measured in kg during study period
Change from baseline in clinical laboratory tests | From Day1 to end-of-study visit (Day 26-28)
  Change from baseline to each time point of measurement during study period for clinical laboratory tests (hematology, clinical chemistry, serology)
Incidence rate of treatment-emergent treatment-emergent adverse events (AEs) and serious adverse events (SAEs) | From Day1 to follow-up period (Day46-48)
  Incidence rates of treatment-emergent AEs including abnormalities in ECG variables during each treatment as well as AEs leading to the discontinuation of study treatment. A treatment-emergent AE is any AE temporally associated with the use of a study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Bruderer, PhD, Study Director — Actelion
Locations (1):
- CRS Clinical Research Services Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No